CLINICAL TRIAL: NCT04008758
Title: Evaluation of Efficacy of Recruitment Maneuver Using Lung Ultrasound in Trauma Patients
Brief Title: Recruitment Maneuver Using Lung Ultrasound in Trauma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AJIRB-MED-OBS-19-119
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Recruitment; Trauma
Keywords: recruitment; ultrasound; trauma; pulmonary contusion
MeSH Terms: conditions — Wounds and Injuries | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Randomized prospective trial
  1. st group is sono group using lung ultrasound
  2. nd group is control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sono group (Experimental): Evaluate the participant's lung condition using ultrasound and do recruitment maneuver if it is necessary
  Interventions: Diagnostic Test: Ultrasound
- control group (No Intervention): If participants need recruitment maneuver (decreasing saturation, peak airway pressure > 35 mmHg) by clinical judgement, do recruitment maneuver not using lung ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Evaluate participant's lung condition using ultrasound. Using lung ultrasound scoring, more than 1 point needs recruitment maneuver
  Arms: sono group

SUMMARY:
In trauma patients, the incidence of pulmonary contusion is frequent. Recruit maneuver using lung ultrasound could be improve oxygenation in trauma populatioin, howevere, there is no previous study. The aim of this study is evaluation of the efficacy of lung recruitment using ultrasound in perioperative period in trauma patients.

DETAILED DESCRIPTION:
In trauma patients, the incidence of pulmonary contusion is 17-75%. Pulmonary contusioin leads to atelectasis, lung consolidatioin. Finally it could results acute respiratory distress syndrome.

Lung ultrasound is non-invasive and available in anytime even during surgery. Previous studies showed recruitment maneuver using ultrasound improved postoperative oxygenation in pediatric cardiac surgery. In adults, recruitment maneuver not using ultrasound improved oxygenation after cardiopulmonary bypass. There is no study in adult trauma population.

The aim of this study is evaluation of the efficacy of lung recruitment using ultrasound in perioperative period in trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Who need surgery under general anesthesia due to trauma
* The position of the surgery is supine

Exclusion Criteria:

* Who has been ventilator care before the surgery
* Thoracic surgery
* Who had cardiopulmonary resuscitation
* Who has acute respiratory distress syndrome

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
arterial oxygen partial pressure / fractional inspired oxygen ratio at end of surgery | 2 hours
  = P /F ratio; Smaller value respresents poor outcome Using arterial blood gas analysis the difference between baseline (immediate after intubation) and end of surgery
  : If P/F ratio difference is improved compared to baseline, it means recruitment maneuver is effective

SECONDARY OUTCOMES:
Lung ultrasound score | 2 hours
  Using lung ultrasound, evaluate lung condition in both group at end of surgery Scoring using "lung ultrasound scoring" Scoring range: 0, normal; 1, small loss of aeration; 2, moderate loss of aeration; 4, severe loss of aeration

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No